CLINICAL TRIAL: NCT02769468
Title: Effect of Temperature Probe Placement in Delivery Room on Temperature at the Admission in the Neonatal Intensive Care Unit (NICU) of Premature Infants?
Brief Title: Effect of Probe Placement in Delivery Room on Temperature at the Admission of Premature Infants?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Responsible Party: Principal Investigator, Dr Brahim Bensouda, MD. Assistant Professor, Maisonneuve-Rosemont Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 15052
Record Dates: First submitted 2016-04-28; First posted 2016-05-11 (Estimated); Last update posted 2017-12-19 (Actual); Status verified 2017-12

CONDITIONS: Body Temperature Changes
Keywords: Temperature-Probe Placement-preterm infant-case room
MeSH Terms: conditions — Body Temperature Changes

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- The Back (Active Comparator): The probe is placed lateral from the spine, 1 cm above the intergluteal cleft, and in side position to the flank between the hips and the ribs.
  Interventions: Other: The Back
- Chest (Active Comparator): The probe is placed on the chest, 1 cm above the left nipple.
  Interventions: Other: Chest
- Left Axilla (Active Comparator): The probe is placed deep in the left axilla
  Interventions: Other: Left Axilla

INTERVENTIONS:
Other: The Back
  Arms: The Back
Other: Chest
  Arms: Chest
Other: Left Axilla
  Arms: Left Axilla

SUMMARY:
The aim of the study is to compare the effect of 3 different skin temperature placement probe in the case room on the admission temperature to the NICU in preterm infants. The authors aim to evaluate which placement results in more preterm in the acceptable range (36.5-37 °C).

DETAILED DESCRIPTION:
It's a prospective randomized trial conducted at Maisonneuve Rosemont Hospital, neonatal tertiary center located in Montreal with over 2600 annual deliveries. All pregnant women who are expecting to deliver a preterm infant with gestational between 28 and 35 6/7 weeks will be eligible to be enrolled into the study and informed consent is obtained.

Simple randomization is accomplished by opening a sealed pre-set envelope with group assignment before delivery.

Group 1: The probe is placed lateral from the spine, 1 cm above the intergluteal cleft, and in side position to the flank between the hips and the ribs.

Group 2: The probe is placed on the chest, 1 cm above the left nipple. Group 3: The probe is placed deep in the left axilla

At birth, all the preterm are immediately placed under a radiant warmer and resuscitated as per Neonatal resuscitation program (NRP) guidelines. Application of a skin temperature probe set at 36.5°C, for servo-controlled thermoregulation by 2 minutes of life. Probes will be fixed with an insulated reﬂective water-soluble gel probe.

No changes are made to the routine delivery room management and resuscitation for this study. After initial delivery room management, babies are transported in a heated radiant warmer (Panda) to the NICU.

In the delivery room, when the baby has a skin temperature servo-controlled stable at 36.5° C, the baby is ready to be transferred to NICU. All babies admitted to the NICU are routinely cared for by the attending neonatologist.

Data collection:

The temperature displaced on the servo controlled table is collected when the baby is the NICU just before transfer from the radiant table to the incubator.

The right axillary temperature will be taken by a thermometer.

ELIGIBILITY:
Inclusion criteria:

* Preterm infant with gestational age between 28 and 35 6/7 weeks

Exclusion criteria:

* Infant with severe congenital malformation and those who had sever asphyxia or died in the delivery room and infant born before arrival of NICU team.

Ages: 28 Weeks to 36 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 121 (Actual)
Dates: Start 2015-11; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
The average temperature right axillary. | 1 year
  The average temperature axillary at the admission in the Neonatal intensive care unit.

CONTACTS AND LOCATIONS:
Overall Officials: Brahim Bensouda, MD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Hopital Maisonneuve Rosemont, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No